CLINICAL TRIAL: NCT06139991
Title: A Phase 1, Randomized, Double-blind, Single-dose, Partial Replicate, 3-period Cross-over Study to Assess the Total Systemic Exposure Bioequivalence of Budesonide and Albuterol Delivered by BDA MDI Hydrofluoroolefin (HFO) Compared With BDA MDI (Hydrofluoroalkene) HFA.
Brief Title: Study to Assess the Pharmacokinetic Bioequivalence of Budesonide and Albuterol With an Alternate Propellant Compared to Current Propellant.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: D6933C00001
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Heathy Participants
Keywords: Albuterol; Budesonide; Combination product; Hydrofluoralkene propellant; Hydrofluoroolefin propellant

STUDY DESIGN:
Intervention Model Description: This is a Partial-replicate, 3-period Cross-over study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Since this is a double-blind study, so the investigator, all clinical staff involved in the clinical study, the participants, and the study monitor will remain blinded, unless safety concerns or a regulatory requirement necessitate unblinding.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment sequence ABB (Experimental): Participants will receive Treatment A, followed by Treatment B, followed by Treatment B, all treatments as a single dose, with a washout period of minimum 3 days, but no longer than 7 days, between each study dose administration.
  Interventions: Drug: Treatment A (BDA MDI HFO); Drug: Treatment B (BDA MDI HFA)
- Treatment sequence BBA (Experimental): Participants will receive Treatment B, followed by Treatment B, followed by Treatment A, all treatments as a single dose, with a washout period of minimum 3 days, but no longer than 7 days, between each study dose administration.
  Interventions: Drug: Treatment A (BDA MDI HFO); Drug: Treatment B (BDA MDI HFA)
- Treatment sequence BAB (Experimental): Participants will receive Treatment B, followed by Treatment A, followed by Treatment B, all treatments as a single dose, with a washout period of minimum 3 days, but no longer than 7 days, between each study dose administration.
  Interventions: Drug: Treatment A (BDA MDI HFO); Drug: Treatment B (BDA MDI HFA)

INTERVENTIONS:
Drug: Treatment A (BDA MDI HFO) — Randomized participants will receive Treatment A (BDA MDI HFO) on Day 1 under fasted condition.
Drug: Treatment B (BDA MDI HFA) — Randomized participants will receive Treatment B (BDA MDI HFA) on Day 1 under fasted condition.

SUMMARY:
This study will investigate the Pharmacokinetic (PK) and safety of Budesonide and albuterol (BDA) metered dose inhaler (MDI) HFO and BDA MDI HFA in healthy male and female participants.

DETAILED DESCRIPTION:
Eligible participant will receive 3 single-dose treatments; 2 doses of BDA MDI HFA and 1 dose of BDA MDI HFO.

* Treatment A: 2 inhalations, single dose of BDA MDI HFO 80/90 μg (test formulation)
* Treatment B: 2 inhalations, single dose of BDA MDI HFA 80/90 μg (reference formulation) Participants will be randomly assigned to receive any 1 of the 3 treatment sequences of ABB, BBA or BAB.

The study will comprise of:

* A screening period of maximum 28 days.
* Three Treatment periods will be up to approximately 22 days (including Follow-up).
* A final follow-up calls within 3-7 days after the last dose of study intervention.

Each participant has to be involved in the study for up to 48 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants (of non-childbearing potential) aged 18 to 60 years, inclusive, with suitable veins for cannulation or repeated venipuncture.
* Female participants must have a negative pregnancy test at screening and on admission and must not be lactating.
* Participants with Body mass index between 18 and 30 kg/m^2, inclusive, and weighing between 50 kg and no more than 120 kg inclusive.
* Participants must have a Forced expiratory volume (FEV)1 ≥ 80% of the predicted normal value and an FEV1/FVC> 70% regarding age, height, and ethnicity at the screening visit.
* Participants must demonstrate proper inhalation technique and is able to use an MDI properly after training.

Exclusion Criteria:

* History or presence of gastrointestinal, hepatic or renal disease, or any other clinically significant disease or disorder.
* History of any clinically significant disease or disorder which may either put the participant at risk because of participation in the study or influence the results or the participant's ability to participate in the study.
* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of study drug.
* Any clinically important abnormalities in clinical chemistry, haematology, or urinalysis results at the screening.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, or Human immunodeficiency virus (HIV).
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting electrocardiogram (ECG) and any clinically important abnormalities in the 12 lead ECG.
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 3 months prior to screening.
* Known or suspected history of alcohol or drug abuse.
* Positive screen for drugs of abuse, alcohol, or cotinine at screening.
* History or presence of severe allergy/hypersensitivity.
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of the study drug.
* Use of any prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, mega dose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks or 5 half-lives of the medication, whichever is longer, prior to the first administration of study drug.
* Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
* Excessive intake of caffeine-containing drinks or food.
* Vulnerable participants.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-05-04 (Actual); Study Completion 2024-05-04 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from time 0 to the last quantifiable concentration (AUClast) | Day 1, Day 2 (pre-dose and post-dose)
  The AUClast of budesonide and albuterol will be evaluated to assess the bioequivalence of the total systemic exposure of budesonide and albuterol administered.
Maximum plasma drug concentration (Cmax) | Day 1, Day 2 (pre-dose and post-dose)
  The Cmax of budesonide and albuterol will be evaluated to assess the bioequivalence of the total systemic exposure of budesonide and albuterol administered.

SECONDARY OUTCOMES:
Area under plasma concentration-time curve from time 0 to infinity (AUCinf) | Day 1, Day 2 (pre-dose and post-dose)
  The AUCinf after administration of budesonide and albuterol will be evaluated.
Time to reach maximum observed concentration (Tmax) | Day 1, Day 2 (pre-dose and post-dose)
  The Tmax after administration of budesonide and albuterol will be evaluated.
Terminal elimination half-life (T1/2λz) | Day 1, Day 2 (pre-dose and post-dose)
  The T1/2λz after administration of budesonide and albuterol will be evaluated.
Mean residence time of the unchanged drug in the systemic circulation from zero to infinity (MRT) | Day 1, Day 2 (pre-dose and post-dose)
  The MRT after administration of budesonide and albuterol will be evaluated.
Apparent total body clearance (CL/F) | Day 1, Day 2 (pre-dose and post-dose)
  The CL/F after administration of budesonide and albuterol will be evaluated.
Apparent volume of distribution during the terminal phase (Vz/F) | Day 1, Day 2 (pre-dose and post-dose)
  The Vz/F after administration of budesonide and albuterol will be evaluated.
Ratio Maximum plasma drug concentration (Cmax) | Day 1, Day 2 (pre-dose and post-dose)
  The ratio of Treatment A (test formulation) and Treatment B (reference formulation) Cmax values will be evaluated.
Ratio Area under plasma concentration-time curve from time 0 to infinity (AUCinf) | Day 1, Day 2 (pre-dose and post-dose)
  The ratio of Treatment A (test formulation) and Treatment B (reference formulation) AUCinf values will be evaluated.
Ratio Are under plasma concentration-time curve from time 0 to the last quantifiable concentration (AUClast) | Day 1, Day 2 (pre-dose and post-dose)
  The ratio of Treatment A (test formulation) and Treatment B (reference formulation) AUClast values will be evaluated.
Number of participants with Adverse Events | From Screening (≤ 28 days to Day -2) until Follow-up phone call (within 3 to 7 days post final dose)
  The safety and tolerability of single doses of BDA MDI HFO and BDA MDI HFA will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information
URL: https://vivli.org/